CLINICAL TRIAL: NCT02343848
Title: Physical Activity and Gestational Complications
Acronym: PEDPTB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Shalom Mazaki-Tovi MD, Directore , HR Unit, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1197-14-SMC
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment (Experimental): smart bracelet.
  Interventions: Device: smart bracelet.

INTERVENTIONS:
Device: smart bracelet. — Physical activity will be evaluated using smart bracelet.

SUMMARY:
The association between physical activity and several complication of pregnancy will be evaluated .

DETAILED DESCRIPTION:
The association between physical activity and several complication of pregnancy will be evaluated. Patients with complications of pregnancy will be recruited. Physical activity will be evaluated using questioner or smart bracelet.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women

Exclusion Criteria:

* Non pregnant women

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-07; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Presence of Gestational Complication | 40 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Shalom Mazaki tovi, Ramat Gan, Israel